CLINICAL TRIAL: NCT01571921
Title: Phase 1a: A Randomized, 2-period Cross-over Study to Compare the Bioavailability of Gamma-Delta Tocotrienol (GDT) With That of Tocotrienol Rich Fraction (TRF) in Twelve Healthy Subjects
Brief Title: Gamma-delta Tocotrienol as Potential Maintenance Treatment in Women With Metastatic Breast Cancer
Acronym: GEMM1a
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Malaysia Palm Oil Board (Other Government)
Collaborators: University of Malaya (Other)
Responsible Party: Principal Investigator, Puvaneswari Meganathan, Ms, Malaysia Palm Oil Board
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 896.128
Record Dates: First submitted 2012-03-26; First posted 2012-04-05 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Gamma-Delta Tocotrienol (Experimental)
  Interventions: Dietary Supplement: Gamma-Delta Tocotrienol and Tocotrienol Rich Fraction
- TRF (Active Comparator)
  Interventions: Dietary Supplement: Gamma-Delta Tocotrienol and Tocotrienol Rich Fraction

INTERVENTIONS:
Dietary Supplement: Gamma-Delta Tocotrienol and Tocotrienol Rich Fraction — Single oral TRF or Gamma-Delta Tocotrienol dosage

SUMMARY:
Twelve healthy volunteers who fit the inclusion and exclusion criteria and provide written informed consent to participate in the trial will be recruited to compare the rate and extent of absorption and pharmacokinetics of the newly formulated Gamma-Delta formulation with TRF.

DETAILED DESCRIPTION:
Twelve healthy subjects will be admitted to a clinical study ward on the Day 0. Physical check up and the health status will be confirmed during check in. After fasting for a minimum of 10 hours overnight, each subject will be administered a single dose of TRF or Gamma-Delta after taking a standardized high-fat meal breakfast on Day 1. Thereafter, standard meals will be provided at 4 and 12 hours after dosing. Blood samples (5mL will be taken using an in-dwelling canula placed in the antecubital vein immediately before and at 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 14, and 24 hours after dosing. Subjects will be admitted for 24 hours and discharged after the last blood sampling. During the study, blood pressure and the heart rate will be monitored regularly for safety profile.

After a one week wash out period, subject will return to the ward and be given the other formulation (TRF or GDT) and the same procedures will be repeated. Any adverse events that arise during the treatment will be recorded and followed up till resolution.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged 21-55 years old
* Good health
* No allergy to vitamin E/ palm oil
* No past (within 3 months) / current use of dietary supplements containing vitamin E

Exclusion Criteria:

* History of bleeding tendencies or any condition predisposing to bleeding e.g. thrombocytopenia, abnormal liver function, liver disease (e.g. chronic hepatitis), gastrointestinal ulcers
* Candidate for surgery or had undergone surgery in the past 6 months
* Current or past use (last 3 months) of antithrombotic drugs such as antiplatelets (aspirin, ticlopidine), anticoagulants (heparin, warfarin), thrombolytic agents (streptokinase), etc
* Current or past history of cancer
* Pregnant/ breastfeeding women
* Smokers
* Drug or alcohol abuse
* Hypercholesterolemia
* Chronic conditions such as uncontrolled hypertension, heart disease (ischemic heart disease, heart failure, cardiac arrhythmia), uncontrolled diabetes, HIV infection, or other psychiatric illness/ social situations that might limit adherence to study protocol.
* Unable or unwilling to stop taking vitamins, herbal preparations or nonprescription medications

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-01; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax)of drug | 0 to 24 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Nur Aishah Mohd Taib, Principal Investigator — University of Malaya
Locations (1):
- University Malaya Medical Centre(UMMC), Lembah Pantai,, Kuala Lumpur, Malaysia

REFERENCES:
- [Background] Patel V, Rink C, Gordillo GM, Khanna S, Gnyawali U, Roy S, Shneker B, Ganesh K, Phillips G, More JL, Sarkar A, Kirkpatrick R, Elkhammas EA, Klatte E, Miller M, Firstenberg MS, Chiocca EA, Nesaretnam K, Sen CK. Oral tocotrienols are transported to human tissues and delay the progression of the model for end-stage liver disease score in patients. J Nutr. 2012 Mar;142(3):513-9. doi: 10.3945/jn.111.151902. Epub 2012 Feb 1. PMID 22298568
- [Background] Mahalingam D, Radhakrishnan AK, Amom Z, Ibrahim N, Nesaretnam K. Effects of supplementation with tocotrienol-rich fraction on immune response to tetanus toxoid immunization in normal healthy volunteers. Eur J Clin Nutr. 2011 Jan;65(1):63-9. doi: 10.1038/ejcn.2010.184. Epub 2010 Sep 22. PMID 20859299
- [Background] Zaiden N, Yap WN, Ong S, Xu CH, Teo VH, Chang CP, Zhang XW, Nesaretnam K, Shiba S, Yap YL. Gamma delta tocotrienols reduce hepatic triglyceride synthesis and VLDL secretion. J Atheroscler Thromb. 2010 Oct 27;17(10):1019-32. doi: 10.5551/jat.4911. Epub 2010 Aug 10. PMID 20702976
- [Background] Comitato R, Nesaretnam K, Leoni G, Ambra R, Canali R, Bolli A, Marino M, Virgili F. A novel mechanism of natural vitamin E tocotrienol activity: involvement of ERbeta signal transduction. Am J Physiol Endocrinol Metab. 2009 Aug;297(2):E427-37. doi: 10.1152/ajpendo.00187.2009. Epub 2009 Jun 2. PMID 19491296
- [Background] Weng-Yew W, Selvaduray KR, Ming CH, Nesaretnam K. Suppression of tumor growth by palm tocotrienols via the attenuation of angiogenesis. Nutr Cancer. 2009;61(3):367-73. doi: 10.1080/01635580802582736. PMID 19373610
- [Result] Nesaretnam K, Selvaduray KR, Abdul Razak G, Veerasenan SD, Gomez PA. Effectiveness of tocotrienol-rich fraction combined with tamoxifen in the management of women with early breast cancer: a pilot clinical trial. Breast Cancer Res. 2010;12(5):R81. doi: 10.1186/bcr2726. Epub 2010 Oct 8. PMID 20929592